CLINICAL TRIAL: NCT00517153
Title: A Phase II Randomized Controlled Study of Miglustat in Adult and Juvenile Patients With Niemann-Pick Type C Disease
Brief Title: Miglustat in Niemann-Pick Type C Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Dr. Ruben Giorgino, Actelion
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OGT-918-007
Record Dates: First submitted 2007-08-15; First posted 2007-08-16 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Niemann-Pick Type C Disease
Keywords: Zavesca; miglustat; Niemann-Pick Type C; Actelion
MeSH Terms: conditions — Niemann-Pick Disease, Type C | interventions — miglustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): OGT-918 - Zavesca (miglustat)
  Interventions: Drug: miglustat
- 2 (No Intervention): Standard treatment

INTERVENTIONS:
Drug: miglustat — Patients aged 12 years or more randomised to the treatment group will receive 200 mg OGT 918 three times daily initially for twelve months. An additional sub-study of up to 12 patients aged under 12 years will receive a lower dose of OGT 918 according to their BSA
  Other Names: Zavesca
  Arms: 1

SUMMARY:
This is a phase II randomized controlled study of miglustat in adult and juvenile patients with Niemann-Pick Type C disease. Up to 42 patients will be randomised in a 2:1 ratio to either treatment with miglustat or to a non-treatment group. Both groups will follow an identical visit schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Niemann-Pick Type C disease confirmed by abnormal cholesterol esterification and abnormal filipin staining.
2. Patients who can ingest a capsule.
3. Patients who are above the age of four (4) years of age.

Exclusion Criteria:

1. Patients younger than 18 years who are unable to give informed assent and/or whose legal guardian is unable to provide informed consent.
2. Patients aged 18 and over who cannot provide informed consent and/or whose legal guardian is unable to provide witnessed informed consent.
3. Sexually active and fertile patients who do not agree to use adequate contraception throughout the study and for three months after cessation of OGT 918 treatment.
4. Patients who cannot tolerate the study procedures or who are unable to travel to the study center as required by this protocol.
5. Patients currently undergoing therapy with other investigational agents or patients taking drugs or food supplements which may interfere with gastrointestinal absorption or motility.
6. Patients suffering from clinically significant diarrhea (>3 liquid stools per day for >7 days) without definable cause within 3 months of Screening Visit, or who have a history of significant gastrointestinal disorders.
7. Patients with an intercurrent medical condition that would render them unsuitable for the study e.g. HIV, hepatitis infection.
8. Patients who in the opinion of the Investigator (for whatever reason) are thought to be unsuitable for the study.
9. Patients with an adjusted Creatinine Clearance of less than 70 ml/min/1.73m2 (CrCl <70).
10. Patients younger than four (4) years of age.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2002-01; Primary Completion 2006-09 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoints will be two parameters - Horizontal Saccadic α and Horizontal Saccadic β - which are estimated for each patient from their saccadic eye movement data | Baseline to Month 12

SECONDARY OUTCOMES:
Highest amplitude for which a velocity measurement is obtained | Baseline to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Chiriboga, Assoc. Prof. MD, Principal Investigator — Columbia University